CLINICAL TRIAL: NCT01883531
Title: A Randomised, Multicentre, Double-blind, Placebo-controlled, Crossover Trial Determining the Efficacy of Dry Powder Mannitol in Improving Lung Function in Subjects With Cystic Fibrosis Aged Six to Seventeen Years
Brief Title: Crossover Trial Determining the Efficacy of Dry Powder Mannitol to Improve Lung Function in Subjects Aged 6-17 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DPM-CF-204; 2012-002699-14 (EudraCT Number)
Record Dates: First submitted 2013-06-17; First posted 2013-06-21 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Cystic Fibrosis
Keywords: improving lung function; paediatric and adolescent; FEV1
MeSH Terms: conditions — Cystic Fibrosis | interventions — Mannitol; Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled Placebo (Placebo Comparator): Eight-week treatment period with inhaled placebo b.d.
  Interventions: Drug: Inhaled Placebo
- Inhaled Mannitol (Active Comparator): Eight-week treatment period Inhaled Mannitol 400 mg b.d.
  Interventions: Drug: Inhaled Mannitol

INTERVENTIONS:
Drug: Inhaled Mannitol — Active treatment is inhaled mannitol with a particle size of 3-4 microns
  Other Names: Mannitol; IDPM; Dry Powder Mannitol for Inhalation; Bronchitol
  Arms: Inhaled Mannitol
Drug: Inhaled Placebo — The PLacebo is non respirable mannitol due to the big size particle
  Other Names: Control
  Arms: Inhaled Placebo

SUMMARY:
It is hypothesised that inhaled mannitol 400 mg b.d. will lead to a significant improvement in the absolute change in percentage of predicted FEV1 from baseline following eight-weeks of trial treatment compared to treatment with inhaled placebo b.d.

Any improvement in FEV1 is considered clinically meaningful; however, this trial has set a threshold of 3% for the purposes of determining an appropriate sample size for statistical power whilst retaining trial feasibility in an orphan disease population.

DETAILED DESCRIPTION:
Drug Name: Dry powder mannitol for inhalation Phase: 2 Indication: Paediatric and adolescent cystic fibrosis Trial Centres: Multicentre Sponsor: Pharmaxis Limited, 20 Rodborough Road, Frenchs Forest, NSW 2086 Australia Trial Duration: 27 weeks Number of Subjects: 160 Trial Design: Randomised, multicentre, double-blind, placebo-controlled, crossover Primary Objective: To determine the effect of eight weeks of twice-daily treatment with inhaled dry powder mannitol on lung function (FEV1) in subjects with CF who are aged six to seventeen years Dosage and Administration: Trial drug is to be administered via a dry powder inhaler.

* Mannitol 400 mg b.d. for 8 weeks followed by a 8-week washout followed by placebo b.d. for 8 weeks; or
* Placebo b.d. for 8 weeks followed by a 8-week washout followed by mannitol 400 mg b.d. for 8 weeks.

Statistical Methods:

* The primary and secondary efficacy analyses will be based upon a modified Grizzle model for crossover design. Absolute and relative changes from baseline in percentage of predicted FEV1 and FVC will be analysed. The absolute change in percentage of predicted lung function (FEV1 and FVC) will be the primary focus. Changes in FEF25-75 will also be analysed.
* Safety data will be analysed descriptively (listings and summary tables).

ELIGIBILITY:
Inclusion Criteria: The subject must:

1. Personally provide, or have a legal guardian provide written informed consent to participate in the trial, according to local regulations;
2. rhDNase and maintenance antibiotic use is allowed but treatment must have been established at least 3 months prior to screening. The subject must remain on rhDNase and / or maintenance antibiotics for the duration of the trial. The subject must not commence treatment with rhDNase or maintenance antibiotics during the trial;
3. Have a confirmed diagnosis of cystic fibrosis (sweat test result greater than or equal to 60 mEq/L chloride and/or genotyping showing two identifiable mutations consistent with a diagnosis of cystic fibrosis);
4. Be aged greater than or equal to 6 years and < 18 years;
5. Have a percentage of predicted FEV1 of greater than or equal to 30% and less than or equal to 90% at Screening (Visit 0). Percentage of predicted FEV1 will be calculated using Wang for children aged < 8 years, and using NHanes III for those greater than or equal to 8 years; and
6. Be able to perform all the techniques necessary to measure lung function.

Exclusion Criteria: The subject must NOT:

1. Be using maintenance nebulised hypertonic saline;
2. Be considered "terminally ill"; eligible for lung transplantation, or have received a lung transplant previously;
3. Require home oxygen or assisted ventilation;
4. Have had an episode of massive haemoptysis defined as acute bleeding ≥240 ml in a 24-hour period and/or recurrent bleeding ≥100 ml/day over several days in the three-months prior to Screening (Visit 0);
5. Have a known intolerance to mannitol;
6. Be taking non-selective beta-blockers;
7. In the three months prior to Screening (Visit 0) have had a myocardial infarction; a cerebral vascular accident; major ocular, abdominal, chest or brain surgery;
8. Have a known cerebral, aortic or abdominal aneurysm;
9. Be currently participating in, or have participated in another investigative drug trial within four weeks of Screening (Visit 0);
10. Be pregnant or breastfeeding, or plan to become pregnant whilst in the trial;
11. For females of childbearing potential, be using an unreliable form of contraception, (at the discretion of the investigator);
12. Have any concomitant medical, psychiatric, or social condition that, in the Investigator's opinion, would put the subject at significant risk, may confound the results or may significantly interfere with the subject's participation in the trial; or
13. Have a "failed" or "incomplete" mannitol tolerance test (as described in Section 8.3.1.1).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2013-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Effect on lung function (FEV1) | The absolute change from each treatment period baseline to week 8 of each treatment period in percentage of predicted FEV1.
  To determine the effect of eight weeks of twice-daily treatment with inhaled dry powder mannitol on lung function (FEV1) in subjects with CF who are aged six to seventeen years.

SECONDARY OUTCOMES:
Effect on FVC | The absolute change from each treatment period baseline to week 8 of each treatment period in percentage of predicted FVC.
  To determine the effect of inhaled mannitol on FVC
Effect of inhaled mannitol on FEF25-75 | The absolute change from each treatment period baseline to week 8 of each treatment period in percentage of predicted FEF25-75.
  To determine the effect of inhaled mannitol on FEF25-75 (exploratory endpoint)
Assess safety | From each treatment period baseline to week 8 of each treatment period.
  Assessment of safety will be made on the basis of reviewing changes in physical examination and using adverse event data.
Sputum weight | The absolute change from each treatment period baseline to week 8 of each treatment period in sputum weight.
  To evaluate the difference in treatment induced sputum weight in subjects treated with inhaled mannitol compared with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Christiane De Boeck, Principal Investigator — UZ Leuven, Belgium; Jeremy Hull, Dr, Principal Investigator — John Radcliffe Hospital, Oxford, UK; Anne Munck, Dr, Principal Investigator — Hôpital Robert Debré, France; Joachim Riethmuller, Dr, Principal Investigator — Universitats Kinderklinik Tubingen, Germany; Larry Lands, MD, Principal Investigator — 'Montreal Children's Hospital, Montreal, Canada; Alexander Möller, MD, Principal Investigator — University Childrens Hospital Zurich; Sonia Volpi, MD, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona Italy; Harm Tiddens, MD, Principal Investigator — Erasmus MC-Sophia Children's Hospital, Rotterdam, Netherlands
Locations (1):
- John Radcliffe Hospital, Oxford, Oxford, United Kingdom